CLINICAL TRIAL: NCT01280227
Title: Supporting Patient Provider Communication for Children With Cancer and Congenital Heart Disease
Brief Title: Supporting Patient Provider Communication in Paediatric Care
Acronym: SiSom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Cornelia Ruland, Professor, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S-05288; 175389/V50
Record Dates: First submitted 2009-09-01; First posted 2011-01-20 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Cancer; Congenital Heart Disease
Keywords: Symptom management; Symptom assessment; Patient satisfaction; Patient-provider communication
MeSH Terms: conditions — Neoplasms; Heart Defects, Congenital; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients uses the symptom assessment tool SiSom. A summary of their reported symptoms are printed out and given to the pediatrician and nurse before the consultation. The consultation is videotaped.
  Interventions: Behavioral: SiSom
- 2 (No Intervention): The control group do not use the symptom assessment tool "SiSom" before the consultation. The control group receives usual care and the consultation is videoptaped.

INTERVENTIONS:
Behavioral: SiSom — SiSom is a symptom assessment tool designed to help the child report disease specific problems.The child also report the severity of their problems. After using the tool a report is printed and given to the clinician.
  Other Names: Symptom assessment tool
  Arms: 1

SUMMARY:
Children with Cancer or congenital heart disease (CHD) experience complex, physical, psychosocial and behavioural symptoms and problems due to the illness, treatment, and medical procedures. To help children cope with their problems and prevent psychological distress, the investigators developed SiSom, a support system to help children with cancer or CHD report their symptoms and problems in an age-adjusted manner on a touch-pad, portable computer.

This quasi-experimental study with 202 children age 7-12 with CHD or cancer will test the following hypotheses: When children use SiSom to report their symptoms and problems, and this information is provided to their clinicians in their outpatient consultations:

* Children and parents will experience less anxiety.
* Children and parents will be more satisfied with the outpatient visit.
* There will be greater congruence between children's reported symptoms and problems and those addressed by their clinicians as evidenced in documented patient care.

To better understand the mechanisms by which these effects may occur, the investigators will also explore:

* Differences between control and experimental groups in patient-provider communication in terms of instrumental and affective behaviour, participation, initiative and person addressed;
* The relationships among outcomes of patient-provider communication, congruence between patients' reported symptoms and those addressed by their clinicians and children's and parents' anxiety and satisfaction; and how these relationships differ between treatment and control conditions.

Finally, the investigators will investigate time requirements, ease of use and usefulness of SiSom by children and clinicians.

For analyses the investigators will use inferential statistics and qualitative analyses of the video-taped consultation sessions. This study will contribute to improving patient-centred care for a particularly vulnerable population, and to a better understanding of the triadic communication and interactions among child-parent and clinician.

ELIGIBILITY:
Inclusion Criteria:

* Between 7 and 12 years.
* Ethnic norwegian.
* Undergoing treatment for cancer or diagnosed with a congenital heart disease.

Exclusion Criteria:

* Receiving or have received radiation the brain as this may affect their abilities to use SiSom and communicate during consultations.
* Syndromes, mental retardation, developmental disorders, language disorders, or cognitive disorders that affect their ability to report symptoms or communicate during consultations.
* Other ethnic origin.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2005-01; Primary Completion 2010-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Patient-provider communication | Single measure, video recording of medical consultation lasting approximately one hour

SECONDARY OUTCOMES:
Patient-provider communication | Single measure, video recording of medical consultation lasting approximately one hour
Time requirements, ease of use | Single measure, after collection of all patient data
Congruence between children's reported symptoms and problems and those addressed by their clinicians as evidenced in documented patient care. | Single measure, ten minutes post intervention
State anxiety | 10 minutes pre and 10 minutes post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia M Ruland, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet-Radiumhospitalet, Oslo, Norway

REFERENCES:
- [Background] Vatne TM, Finset A, Ornes K, Ruland CM. Application of the verona coding definitions of emotional sequences (VR-CoDES) on a pediatric data set. Patient Educ Couns. 2010 Sep;80(3):399-404. doi: 10.1016/j.pec.2010.06.026. PMID 20663629
- [Background] Ruland CM, Starren J, Vatne TM. Participatory design with children in the development of a support system for patient-centered care in pediatric oncology. J Biomed Inform. 2008 Aug;41(4):624-35. doi: 10.1016/j.jbi.2007.10.004. Epub 2007 Nov 13. PMID 18082468
- [Background] Ruland CM, Slaughter L, Starren J, Vatne TM, Moe EY. Children's contributions to designing a communication tool for children with cancer. Stud Health Technol Inform. 2007;129(Pt 2):977-82. PMID 17911861
- [Background] Slaughter LA, Ruland CM, Vatne TM. Constructing an effective information architecture for a pediatric cancer symptom assessment tool. AMIA Annu Symp Proc. 2006;2006:1102. PMID 17238721
- [Background] Ruland CM, Slaughter L, Starren J, Vatne TM. Children as design partners in the development of a support system for children with cancer. Stud Health Technol Inform. 2006;122:80-5. PMID 17102222
- [Result] Vatne TM, Ruland CM, Ornes K, Finset A. Children's expressions of negative emotions and adults' responses during routine cardiac consultations. J Pediatr Psychol. 2012 Mar;37(2):232-40. doi: 10.1093/jpepsy/jsr074. Epub 2011 Sep 9. PMID 21908544
- [Result] Vatne TM, Slaugther L, Ruland CM. How children with cancer communicate and think about symptoms. J Pediatr Oncol Nurs. 2010 Jan-Feb;27(1):24-32. doi: 10.1177/1043454209349358. Epub 2009 Oct 15. PMID 19833978